CLINICAL TRIAL: NCT05301595
Title: Transversus Abdominus Plane Block Versus Quadratus Lumborum Block for Postoperative Analgesia After Abdominal-based Free Tissue Transfer for Breast Reconstruction After Mastectomy
Brief Title: TAP vs QL for Postoperative Analgesia After DIEP Free Flap Breast Reconstruction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was never started as PI moved to another city
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Moein Momtazi, Plastic and Reconstructive Surgeon, Ottawa Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20210817-01H
Record Dates: First submitted 2022-03-08; First posted 2022-03-29 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will be randomized to receive intraoperative TAP block (Group A) or preoperative ultrasound- guided QL block (Group B).
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients will be randomized by using forty-six sealed, opaque envelopes to receive a TAP block or QL block.
  This is a double-blind study. Patient, surgeon and study staff will know which group patient has been assigned to. The anesthetist will know which group you are in for logistical purposes. The patient and surgeon will not know which nerve block the patient received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP block (Active Comparator): All patients will have paravertebral (PV) blocks of the chest performed prior to induction of general anesthesia.
  Patients in this group will have bilateral sham blocks performed after PV block is complete. 2ml of normal saline will be injected under the skin bilaterally near the insertion site of a typical QL block.
  TAP block will be performed intraoperatively by the surgeon. The anesthesiologist will provide the surgeon with 40ml of LA mixture (ropivacaine 0.25%, epinephrine 100mcg and dexamethasone 4mg) for patients in this group. The surgeon will be blinded to the injectate content. The TAP block is performed once the abdominal flap has been harvested. The triangle of Petit is landmarked by the iliac crest inferiorly, the latissimus dorsi muscle posteriorly and the external oblique muscle anteriorly. A blunt tip needle is advanced through the external oblique fascia and internal oblique fascia. A total volume 20mL of the LA mixture will be injected per side.
  Interventions: Procedure: TAP block
- QL block (Active Comparator): All patients will have paravertebral (PV) blocks of the chest performed prior to induction of general anesthesia.
  Patients in this group will have QL block performed after PV block is complete. This will be performed with patients in the prone position using the transverse in-plane technique. With realtime U/S guidance, the quadratus lumborum muscle is identified before a short-bevel needle is advanced into the plane between the quadratus lumborum and psoas major muscles. Needle tip position is confirmed by separation of quadratus lumborum and psoas major upon injection. 20ml of ropivacaine 0.25%, epinephrine 50mcg and dexamethasone 2mg will be injected per side.
  TAP block is performed intraoperatively similar to above but with 40mL of normal saline to perform a sham block. The anesthesiologist will provide the surgeon with 40ml of normal saline in this group. The surgeon will be blinded to the injectate content.
  Interventions: Procedure: QL Block

INTERVENTIONS:
Procedure: TAP block — Please see description of TAP block group.
  Arms: TAP block
Procedure: QL Block — Please see description of QL block group.
  Arms: QL block

SUMMARY:
The purpose of this study is to compare the efficacy of Transversus abdominus plane (TAP) block and Quadratus Lumborum (QL) block on the quality of recovery after breast reconstruction with deep inferior epigastric perforator (DIEP) flap.

DETAILED DESCRIPTION:
Breast reconstruction after mastectomy has seen continued growth and popularity in recent years secondary to improved surgical techniques and improved patient awareness and understanding. While implant-based reconstruction remain the most popular option, autologous tissue transfer, reconstruction of the breast with a patient's own tissues, has emerged as the gold standard for breast reconstruction, most commonly performed with abdominally-based flaps, such as the deep inferior epigastric perforator (DIEP) flap.

Postoperative pain can be a difficult challenge in patients who have undergone DIEP flap. Patients with worse postoperative pain control report worse overall satisfaction with their surgical experience.

A multimodal analgesia protocol is a key component in the postoperative care after DIEP flap. Regional nerve blocks present an adjunct to these protocols that can potentially improve the quality of recovery of these patients.

Transversus abdominus plane (TAP) blocks have been shown to be a safe and effective technique to manage postoperative pain at the abdomen in this population; lowering usage of opiates, shortening length of stay and reducing episodes of nausea and vomiting. TAP's efficacy is well-established and documented for postoperative analgesia in abdominal surgery. This can be done preoperatively by an anesthetist via ultrasound-guidance or, using traditional technique of direct visualization, intraoperatively by the operating surgeon. Surgeon-performed intra-operative TAP block are often preferred as it is less time-consuming. TAP block has become the standard abdominal regional nerve block to perform during this procedure.

More recently, QL block has emerged as an alternative to TAP block for lower abdominal surgery. The QL block is an ultrasound-guided fascial plane block performed by an anesthetist for anterior abdominal wall analgesia.

This study will compare QL block to TAP block in patients undergoing DIEP free flap breast reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* Women (age 18 years or older) who are booked for abdominally based free flap for breast reconstruction
* Patients with America Society of Anesthesiologists (ASA) physical status class I, II and III

Exclusion Criteria:

* Patients not consenting for regional block
* Patients allergic to local anesthetics and adjuvants
* Patients with America Society of Anesthesiologists (ASA) physical status class IV and V
* Patients with any baseline opiate consumption
* Presence of infection at needle insertion site
* Patients with coagulopathy (INR>1.3)
* Patients with thrombocytopenia (Platelets<100)
* Patients on therapeutic anticoagulation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-04 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery-15 survey | post-operative day #1
  Quality of Recovery-15 (QoR-15) survey is a validated 15-item patient-rated postoperative recovery score, will be obtained on postoperative day (POD) 1. Survey results are a numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery). Higher scores are a better outcome.

SECONDARY OUTCOMES:
Quality of Recovery-15 survey | post-operative day #2
  Quality of Recovery-15 (QoR-15) survey is a validated 15-item patient-rated postoperative recovery score, will be obtained on postoperative day (POD) 2. Survey results are a numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery). Higher scores are a better outcome.
Quality of Recovery-15 survey | post-operative day #3
  Quality of Recovery-15 (QoR-15) survey is a validated 15-item patient-rated postoperative recovery score, will be obtained on postoperative day (POD) 3. Survey results are a numerical rating scale leads to a minimum score of 0 (very poor recovery) and a maximum score of 150 (excellent recovery). Higher scores are a better outcome.
Pain visual analog scale | 1st, 2nd, 4th, 8th, 12th, 16th and 24th postoperative hours
  Pain visual analog scale (VAS) is a 1 to 10 continuous scale used to determine the intensity of a patient's pain at any given time. For any given time, the minimum value is 1 (no pain) and the maximum value is 10 (pain as bad as it could possibly be). The lower the number, the less intense the pain and better outcome.
Time elapsed before first analgesic requirement | post-operative day #0 to 3
  Time that has elapsed since surgery before first analgesic medication is needed.
Total analgesic drug requirements | post-operative day #0 to 3
  The total amount of analgesic medication patient requires in the first 3 days after surgery
Total antiemetic drug requirements | post-operative day #0 to 3
  The total amount of antiemetic medication patient requires in the first 3 days after surgery
Ambulation | post-operative day #0 to 3
  Ability of patient to ambulate (e.g. up to chair, mobilizing with assistance, mobilizing independently) in the first 3 days after surgery.
Surgical complication | post-operative day #0 to 3
  Any acute surgical complications experienced by the patient in the first three days after surgery.
Block complication | post-operative day #0 to 3
  Any acute nerve-block related complications experienced by the patient in the first three days after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Moein Momtazi, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No